CLINICAL TRIAL: NCT05454137
Title: Postural Orthostatic Tachycardia Syndrome: a Pilot, Feasibility Study of an Integrative Shared Medical Appointment Intervention
Brief Title: A Shared Medical Appointment Intervention for Quality of Life Improvement in POTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001552
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-12

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Shared Medical Appointments

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- participate in shared medical appointment (Experimental): The POTS shared medical appointment will occur once monthly for four months. Each visit will last 1.5 hours. The group will meet in our clinic group space and lifestyle management therapies will be taught by a physician and another provider ie occupational therapist, dietician etc
  Interventions: Behavioral: Shared medical appointment
- Do not participate in shared medical appointment (No Intervention): participants will only have one-on-one traditional visit with the physician

INTERVENTIONS:
Behavioral: Shared medical appointment — Shared medical appointment
  Arms: participate in shared medical appointment

SUMMARY:
Postural orthostatic tachycardia syndrome (POTS) is a clinical syndrome encompassing a myriad of debilitating symptoms that does not have any FDA approved drug therapies. We propose a shared medical appointment intervention where participants will learn lifestyle management therapies and integrative practices that may improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patients with a physician diagnosis of POTS

Exclusion Criteria:

* patients with uncontrolled psychiatric disease
* patients with uncontrolled medical illness including recent myocardial infarction, stroke, and active malignancy
* non-English speakers as the group intervention will be delivered in English
* pregnant women

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention rate | at 4 months
  Percentage of participants who consent to study participation, attend sessions, and complete the program and scheduled outcome assessments

SECONDARY OUTCOMES:
Change in COMPASS overall score | Baseline and 4 months
  The Composite Autonomic Symptom Score is a self-assessment of autonomic function: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor.
Change on Short Form Survey (SF-36) overall score | Baseline and 4 months
  The 36-Item Short Form Survey (SF-36), is a self assessment of vitality, physical functioning, bodily pain, health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health

CONTACTS AND LOCATIONS:
Overall Officials: Talal Moukabary, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No